CLINICAL TRIAL: NCT02620891
Title: Study on the Effect of Helium Oxygen Mixture in the Treatment of Meconium Aspiration Syndrome Parallel Synchronized Intermittent Mandatory Ventilation; Synchronous Maudatory Ventilation
Brief Title: Helium Oxygen Mixture in the Treatment of Meconium Aspiration Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ma Juan (Other)
Responsible Party: Sponsor-Investigator, Ma Juan, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Organization: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MJuan
Record Dates: First submitted 2015-11-12; First posted 2015-12-03 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Neonatal Meconium Aspiration
Keywords: helium oxygen mixture; Meconium aspiration syndrome
MeSH Terms: conditions — Meconium Aspiration Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group (Active Comparator): Using helium oxygen mixture
  Interventions: Device: helium oxygen mixture
- matched group (No Intervention): Using air oxygen mixture

INTERVENTIONS:
Device: helium oxygen mixture
  Other Names: Air oxygen mixture
  Arms: experimental group

SUMMARY:
Helium-oxygen mixture(heliox) was suggested to be beneficial in meconium aspiration syndrome in previous studies，but the evidence was limited．The aim of the study was to assess the effectiveness of synchronize intermittent mandatory ventilation (SIMV) with heliox (70% helium and 30% oxygen) on length of ventilation(LoV) and cardiopulmonary protection in meconium aspiration syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Subject has the diagnosis of neonatal meconium aspiration syndrome
* Subject has Synchronous instruction ventilation

Exclusion Criteria:

* History of congenital or hereditary disease

Ages: 37 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
blood gas analysis | 2 hour
  Time detection after treatment
blood gas analysis | 6 hour
blood gas analysis | 12 hour
blood gas analysis | 24 hour
blood gas analysis | 48 hour

SECONDARY OUTCOMES:
Inflammatory response index (IL-6,IL-8, TNF-a,CRP) | 0 hour
Inflammatory response index (IL-6,IL-8, TNF-a,CRP) | 6 hour

OTHER OUTCOMES:
Amplitude integrated electroencephalogram | 28and 100 days
Amplitude integrated electroencephalogram | 100 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China